CLINICAL TRIAL: NCT04674566
Title: Randomized, Double-blind, Placebo Controlled, Parallel Group, Multi-centre, First-in-human, Phase Ib/II Study to Assess Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, Immunogenicity, and Efficacy of COR-101 in Hospitalized Patients
Brief Title: Evaluation of Safety and Tolerability of COR-101 in Hospitalized Patients With Moderate to Severe COVID-19
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Corat Therapeutics Gmbh (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COR-101/001
Record Dates: First submitted 2020-12-17; First posted 2020-12-19 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): COR-101 low dose
  Interventions: Drug: COR-101; Drug: Placebo
- Cohort 2 (Experimental): COR-101 mid dose 1
  Interventions: Drug: COR-101; Drug: Placebo
- Cohort 3 (Experimental): COR-101 mid dose 2
  Interventions: Drug: COR-101; Drug: Placebo
- Cohort 4 (Experimental): COR-101 high dose
  Interventions: Drug: COR-101; Drug: Placebo

INTERVENTIONS:
Drug: COR-101 — Administered intravenously (IV) single dose
Drug: Placebo — Administered intravenously (IV) single dose

SUMMARY:
Primary objectives Part 1:

- To evaluate the safety and tolerability of COR-101 compared to placebo

Secondary objectives Part 1:

* To evaluate the preliminary efficacy of COR-101 compared to placebo in hospitalized patients with moderate to severe COVID-19
* To assess the pharmacokinetics (PK), pharmacodynamics (PD), and immunogenicity of COR-101

ELIGIBILITY:
Key Inclusion Criteria:

* Hospitalized for COVID-19 illness for ≤72 hours
* Positive SARS-CoV-2 test by standard RT-PCR assay or equivalent test
* Presence of moderate to severe clinical signs indicative of moderate or severe illness with COVID19 prior to study treatment

Key Exclusion Criteria:

* Diagnosis of asymptomatic COVID-19, mild COVID-19, or critical COVID-19
* In the opinion of the investigator, is not likely to survive for >48 hours beyond Day 1
* New onset stroke or seizure disorder during hospitalization and prior to Day 1
* History of relevant CNS pathology or current relevant CNS pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-04-21 (Actual); Primary Completion 2022-10-30 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with Treatment-Emergent Adverse Events (TEAEs) | through Day 28
Proportion of patients with Serious Adverse Events (SAEs) | through Day 28
Proportion of patients with Adverse Events of Special Interest (AESI) | through Day 28

SECONDARY OUTCOMES:
Secondary efficacy endpoint: Proportion of patients with disease progression | through Day 28
  Proportion of patients who are not alive or have respiratory failure
Secondary efficacy endpoint: Time to negative RT-PCR for SARS-CoV-2 | through Day 28
Assessment of pharmacokinetic (PK) parameter: maximum serum concentration observed (Cmax) of COR-101 | through Day 60
Assessment of PK parameter: Time to Cmax (tmax) for COR-101 | through Day 60
Assessment of PK parameter: AUC from time zero extrapolated to infinity (AUCinf) for COR-101 | through Day 60
Assessment of PK parameter: Clearance (CL) for COR-101 | through Day 60
Assessment of PK parameter: Mean residence time (MRT) of COR-101 | through Day 60
Secondary PD endpoint: Change of the viral load of SARS-CoV-2 from baseline, as measured from nasopharyngeal swab samples by qRT-PCR | through Day 21
Secondary immunogenicity endpoint: Percentage of patients with detectable neutralizing antibodies to COR-101 | through Day 60

CONTACTS AND LOCATIONS:
Overall Officials: Helmut Salih, Principal Investigator — University Hospital Tübingen
Locations (1):
- University Hospital Tübingen, Tübingen, Germany

REFERENCES:
- [Derived] Marconato M, Hackenbruch C, Jager S, Gopel S, capital KA, Cyrillicirieieva T, Gavrylov A, Fricke H, Hust M, Dubel S, Dings C, Lehr T, Cuevas M, Bitzer M, Klein C, Schwab M, Wirtz H, Schneider J, Bitter T, Frenzel A, Dhaen MA, Herrmann A, Jung G, Walz JS, Salih HR, Heitmann JS. Phase I Study Evaluating a Monoclonal Fc-Silenced SARS-CoV-2 Antibody in Patients With Moderate-to-Severe COVID-19. Clin Ther. 2026 Feb 6:S0149-2918(26)00007-X. doi: 10.1016/j.clinthera.2026.01.004. Online ahead of print. PMID 41654452
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343